CLINICAL TRIAL: NCT03929510
Title: A PHASE 1, OPEN-LABEL, NON-RANDOMIZED, 2-PERIOD, FIXED SEQUENCE STUDY TO INVESTIGATE THE ABSORPTION, DISTRIBUTION, METABOLISM AND EXCRETION OF 14C-PF-06651600 AND TO ASSESS THE ABSOLUTE BIOAVAILABILITY AND FRACTION ABSORBED OF PF-06651600 IN HEALTHY MALE PARTICIPANTS USING A 14C-MICROTRACER APPROACH
Brief Title: Study to Characterize Absorption, Distribution, Metabolism and Excretion of 14C PF-06651600 and to Evaluate the Absolute Oral Bioavailability and Fraction Absorbed of PF-06651600.
Acronym: B7981011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: B7981011; 2018-003551-38 (EudraCT Number)
Record Dates: First submitted 2019-04-17; First posted 2019-04-29 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; Male; healthy
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Period A (Experimental): Single oral dose of 200 mg 14C labeled PF-06651600 containing approximately 300 nCi 14C (ie, radiolabeled PF 06651600).
  Interventions: Drug: 14C-PF-06651600
- Period B (Experimental): Single oral dose of 200 milligrams (mg) unlabeled PF-06651600 followed at time of peak plasma concentration (Tmax) by an Intravenous (IV) dose of 60 micrograms.14C -PF-06651600 containing approximately 300 nCi 14C (ie, radiolabeled PF-06651600).
  Interventions: Drug: 14C-PF-06651600 IV; Drug: PF-06651600

INTERVENTIONS:
Drug: 14C-PF-06651600 — Oral solution of 200 mg 14C labeled PF-06651600 containing approximately 300 nCi radioactivity
  Arms: Period A
Drug: 14C-PF-06651600 IV — IV solution 60 micrograms of 14C labeled PF-06651600 containing approximately 300 nCi radioactivity
  Arms: Period B
Drug: PF-06651600 — Oral solution 200mg
  Arms: Period B

SUMMARY:
This study will investigate the absorption, distribution, metabolism and excretion (ADME) of 14C PF-06651600 and characterize plasma, fecal and urinary radioactivity and identify any metabolites, if possible, of 14C PF-06651600 in humans.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are healthy as determined by medical evaluation including a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate (PR) measurement, 12 lead ECG, and clinical laboratory tests.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Known immunodeficiency disorder, including positive serology for human immunodeficiency virus (HIV) at screening, or a first degree relative with a hereditary immunodeficiency.
* Infection with hepatitis B or hepatitis C viruses.
* Participants with selected acute or chronic infections or infection history.
* Participants have a known present or a history of malignancy other than a successfully treated or excised non metastatic basal cell or squamous cell cancer of the skin.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
* Use of tobacco/nicotine containing products within 3 months prior to dosing or positive urine cotinine test.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only Male participants will be enrolled.
Enrollment: 6 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Mass Balance: Cumulative recovery (%) of radioactivity in urine | from time zero to the time of last measurable concentration following oral administration of 14C PF-06651600 microtracer dose up to day 24
  Cumulative recovery (%) of radioactivity in urine.
Mass Balance: Cumulative recovery (%) of radioactivity in feces | from time zero to the time of last measurable concentration following oral administration of 14C PF-06651600 microtracer dose up to day 24
  Cumulative recovery (%) of radioactivity in feces

SECONDARY OUTCOMES:
Amount (% of the administered dose) of major metabolites of PF-06651600 in plasma | Hour 0 up to 312 hours post-dose.
Amount (% of the administered dose) of major metabolites of PF-06651600 in urine | Hour 0 up to 312 hours post-dose.
Amount (% of the administered dose) of major metabolites of PF-06651600 in feces | Hour 0 up to 312 hours post-dose.
Cmax | Pre-dose, 0.25. 0.5, 1, 1.5, 2, 3.5, 4.5, 6.5, 8.5, 12.5, 24, 48, 72, 96 hours post-dose
  Maximum plasma concentration
AUClast | Pre-dose, 0.25. 0.5, 1, 1.5, 2, 3.5, 4.5, 6.5, 8.5, 12.5, 24, 48, 72, 96 hours post-dose
  Area under the plasma concentration time profile from time 0 to time of the last quantifiable concentration (Clast)
AUCinf | Pre-dose, 0.25. 0.5, 1, 1.5, 2, 3.5, 4.5, 6.5, 8.5, 12.5, 24, 48, 72, 96 hours post-dose
  Area under the plasma concentration time profile from time 0 to infinity
Tmax | Pre-dose, 0.25. 0.5, 1, 1.5, 2, 3.5, 4.5, 6.5, 8.5, 12.5, 24, 48, 72, 96 hours post-dose
  Time for Cmax
t1/2 | Pre-dose, 0.25. 0.5, 1, 1.5, 2, 3.5, 4.5, 6.5, 8.5, 12.5, 24, 48, 72, 96 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
CL (IV) | Pre-dose, 0.25. 0.5, 1, 1.5, 2, 3.5, 4.5, 6.5, 8.5, 12.5, 24, 48, 72, 96 hours post-dose
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes). Clearance obtained after intravenous infusion dose (apparent clearance) is influenced by the fraction of the dose absorbed.
CL/F (oral) | Pre-dose, 0.25. 0.5, 1, 1.5, 2, 3.5, 4.5, 6.5, 8.5, 12.5, 24, 48, 72, 96 hours post-dose
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes). Clearance obtained after intravenous infusion dose (apparent clearance) is influenced by the fraction of the dose absorbed.
Vss | Pre-dose, 0.25. 0.5, 1, 1.5, 2, 3.5, 4.5, 6.5, 8.5, 12.5, 24, 48, 72, 96 hours post-dose
  Steady state volume of distribution following IV infusion
Vz/F | Pre-dose, 0.25. 0.5, 1, 1.5, 2, 3.5, 4.5, 6.5, 8.5, 12.5, 24, 48, 72, 96 hours post-dose
  Apparent volume of distribution following oral administration
Total 14C_Urine_PO | Pre-dose, Day1, day 2, day 3, day 4, day 5, day 6 and day 7 post-dose
  Total radioactivity excreted into the urine from time zero to the time of last measurable concentration following oral administration of 14C PF 06651600 microtracer dose
Total 14C_Urine_IV | Pre-dose, Day1, day 2, day 3, day 4, day 5, day 6 and day 7 post-dose
  Total radioactivity excreted into the urine from time zero to the time of last measurable concentration following IV administration of 14C PF 06651600 microtracer dose
AE | Baseline (Day 0) up to 90 days after last dose of study medication
  Number of subjects and number of AEs which are any untoward medical occurrence regardless of attribution to study drug in a participant who received study drug.
Number of participants with clinically significant changes to the physical examination | Baseline (Day 0) up to Day 24
  clinically significant changes to the physical examination
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline (Day 0) up to Day 24
  Vital signs (temperature, respiratory rate, pulse, systolic and diastolic blood pressure) obtained from each participant. Clinical significance of vital signs was determined at the investigator's discretion.
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline (Day 0) up to Day 24
  Laboratory parameters include: hematological and chemical parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Netherlands (2):
  - PRA Health Sciences, Groningen
  - PRA Health Sciences Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7981011&StudyName=A+Phase+1%2C+Open-label%2C+Non-randomized%2C+2-period%2C+Fixed+Sequence+Study+To+Investigate+The+Absorption%2C+Distribution%2C+Metabolism+And+Excretion+Of+14c-pf-06651600+And+To+Assess+The+Absolute+Bioavailability+And+Fraction+Absorbed+Of+Pf-06651600+In+Healthy+Male+Participants+Using+A+14c-microtracer+Approach